CLINICAL TRIAL: NCT00295282
Title: A Phase I, Multicenter, Dose-escalation Study of MDX-1100 (Anti-CXCL10 Human Monoclonal Antibody) in Patients With Active Ulcerative Colitis
Brief Title: A Dose-Escalation Study of MDX-1100 in Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX1100-01; IM129-001 (Other: BMS)
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; UC; Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Colitis | interventions — MDX-1100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): patients will receive active MDX-1100
  Interventions: Drug: MDX-1100 (anti-CXCL10 human monoclonal antibody)

INTERVENTIONS:
Drug: MDX-1100 (anti-CXCL10 human monoclonal antibody) — Patients will receive a single dose of MDX-1100 at 0.3, 1.0, 3.0 or 10 mg/kg as a 60 minute intravenous infusion. Patients who respond to treatment may receive up to an additional 3 doses of MDX-1100.

SUMMARY:
This is a Phase I dose-escalation study of MDX-1100. patients with ulcerative colitis will be enrolled into one of four dose cohorts, to receive of MDX-1100 at 0.3, 1.0, 3.0 or 10mg/kg. Three to six patients will be enrolled at each dose level, starting at the lowest dose level, for a maximum of 24 patients to be enrolled into the study. The study is designed to establish the safety and tolerability of single doses of MDX-1100 administered in dose-escalating cohorts to patients with ulcerative colitis. Other study objectives include characterizing a pharmacokinetic profile and pharmacodynamic effects of MDX-1100 and determination of immunogenic response to MDX-1100.

DETAILED DESCRIPTION:
The primary objectives of this study is to establish the safety and tolerability of single doses of MDX-1100 administered in dose-escalating cohorts to patients with active ulcerative colitis (UC).

The secondary objectives include:

1. to characterize the pharmacokinetic profile of MDX-1100,
2. to determine the pharmacodynamic effects of MDX-1100 on CXCL10-related surrogate markers,
3. to obtain preliminary evidence as assessed by the Ulcerative Colitis Disease Activity Index (DAI),
4. to determine the immunogenic response to MDX-1100, and
5. determine the safety and efficacy of repeat doses in patients who respond to a single dose of MDX-1100.

This is a Phase I, multicenter, dose-escalation study of MDX-1100 (anti-CXCL10 human monoclonal antibody) in patients with UC, as defined by standard clinical, endoscopic and histological criteria and a DAI greater than or equal to 4 and less than or equal to 9. Three to six patients will be entered into each of 4 cohorts (0.3, 1.0, 3.0 or 10mg/kg). Starting with the lowest dose cohort (0.3mg/kg), patients will be administered a single dose of MDX-1100 at Day 1 and will be followed until 70 days from the last dose. Dose escalation may proceed when the third patient in the cohort has reached Day 29 and if no dose-limiting toxicities (DLTs) have occurred. Dose escalation may proceed when the sixth patient reaches Day 29 and <2 DLTs have occurred in the cohort. Dose escalation will continue until the last cohort is enrolled or the maximum tolerated dose (MTD) is defined.

Patients who respond to the initial dose, as defined by a decrease in the UC disease activity index (UCDAI) by greater than or equal to 3 points at Day 29 compared to baseline, will be offered the option of receiving up to 3 additional doses of MDX-1100 at their originally assigned dose level. Re-dosing will be permitted at the time of disease flare which is defined as a worsening of the modified UCDAI of greater than or equal to 2 compared to the prior nadir. In order to obtain PK data, the first re-dose may not be administered until Day 43 and all subsequent doses may be great than or equal to 28 days apart. A response in the repeat dosing phase will be defined as a decrease in the mUCDAI of greater than or equal to 2 as compared to the previous baseline mUCDAI. For the second infusion, the comparison will use the mUCDAI calculated at Day 29 or subsequent nadir.

The study will terminate approximately 70 days after the last patient has received the last dose of MDX-1100. It is anticipated that the maximum total time on study for any patient will be less than 1 year.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent and HIPAA
* must be 18 years or older
* patients with active ulcerative colitis with a UCDAI greater than or equal to 4 and less than or equal to 9.
* certain medications initiated at specific schedules prior to study drug administration may be enrolled.
* must meet screening laboratory values
* women of childbearing potential must be using effective contraception for at least 1 month prior to study entry and agree to continue contraception for the duration of their participation in the study, and
* Sexually active male patients must use a barrier method of contraception during the course of the study.

Exclusion Criteria:

* History of colectomy, partial colectomy, current ostomy, or pouchitis
* Presence of Cushing's Syndrome
* Toxic megacolon or fulminant disease likely to require colectomy
* Prior treatment with any monoclonal antibody or immunoglobulin-based fusion proteins 8 weeks or less prior to treatment with MDX-1100
* Any experimental treatment 4 weeks or less prior to treatment with MDX-1100
* Primary or secondary immunodeficiency
* Any history of malignancy, excluding adequately treated and cured basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ
* Active major psychiatric disease(stable depression receiving appropriate medical management will be permitted)
* Evidence of acute or chronic infection or neoplasm on Screening chest radiography
* Current treatment for TB or positive PPD without prophylaxis
* Herpes zoster 3 months or less prior to screening
* Clinically significant cardiac disease requiring medication, unstable angina, myocardial infarction within 6 months, or congestive heart failure
* Active infectious disease requiring i.v. antibiotics within the past 4 weeks or oral antibiotics at the time of enrollment
* Arrhythmia requiring active therapy, with the exception of clinically insignificant extrasystoles, or minor conduction abnormalities
* History of cerebrovascular disease requiring medication/treatment
* Anticoagulation therapy or a known bleeding disorder
* Seizure disorder requiring active therapy
* Known drug or alcohol abuse
* Positive tests for HIV, HBV, or HCV
* Pregnant or nursing
* Any underlying medical condition that in the Investigator's opinion will make the administration of study drug hazardous to the patient or would obscure the interpretation of adverse events, or
* Inability or unwillingness to return for Follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
incidence and severity of treatment-emergent adverse events | events will be followed to resolution

SECONDARY OUTCOMES:
vital sign measurements | study duration - each visit
clinical laboratory tests | study duration - each visit
immunogenicity assessment | dosing and follow up phases
physical examinations | study duration - each visit
Electrocardiograph | periodically through study duration
pharmacokinetic sampling | during dosing phase

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - DMI Health Care Group, Inc., Largo, Florida
  - Metropolitan Gastroenterology Group, PC, Chevy Chase, Maryland
  - University of Medicine and Dentistry of New Jersery (UMDNJ), New Brunswick, New Jersey
  - Mount Sinai School of Medicine, New York, New York